CLINICAL TRIAL: NCT05811130
Title: Examinating Premenstrual Syndrome and Its Influencing Factors Such as Physical Activity, Perceived Stress and Mental Status - Cross Sectional Study
Brief Title: Premenstrual Syndrome and Its Influencing Factors Such as Physical Activity, Perceived Stress and Mental Status
Status: Completed | Type: Observational
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Other Study IDs: 9386/2022
Record Dates: First submitted 2023-03-14; First posted 2023-04-13 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Premenstrual Syndrome
Keywords: physical activity; perceived stress; mental health
MeSH Terms: conditions — Premenstrual Syndrome; Motor Activity; Psychological Well-Being

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our research aimed to investigate how a sedentary lifestyle, body mass index, depression, and stress affect the severity of PMS symptoms and how the listed factors influence each other.

DETAILED DESCRIPTION:
The measuring instrument used was compiled from standard and self-made questionnaires.

The data collection spanned 6 months on the Google Forms platform. The sampling procedure used was convenience sampling. 500 people were invited to fill out the questionnaire, which was sent to women's health-themed groups on social media, and it was also sent to universities in Hungary.

At the same time as the cross-sectional research, the investigators formed two groups concerning the results of the Premenstrual Assessment Form questionnaire: a case group and a control group. The obtained results were examined for both the experimental and control groups.

The self-edited part of the examining tool consisted of general questions (socio-demographic, women's and public health, anthropometric) and standardized questionnaires integrated into the online questionnaire.

The investigators assessed the age of the subjects and calculated their body mass index (BMI) by assessing the participants weight and height.

During the questionnaire, The investigators covered the lifestyle of the subjects: smoking, coffee, alcohol, and drug consumption habits. The investigators asked about the characteristics of the menstrual cycle, such as the presence of pain and cramps or the regularity of the cycle (a cycle between 21-35 days was considered regular). The investigators have also assessed the presence of pregnancy and breastfeeding.

In general questions about physical activity, the investigators collected data on how often subjects engage in physical activity.

The General Health Questionnaire-12

To assess the presence of depression, the investigators used Goldberg's 12-item General Health Questionnaire (GHQ-12). The original questionnaire consisted of 60 questions, and several versions have proven useful over time. The questionnaire assesses mental health through 4 subscales: somatic symptoms, anxiety and insomnia, social dysfunctions, and severe depression. The participants could answer the 12 questions on a scale from 0 to 3. Two scoring systems can be used when evaluating the GHQ-12: the so-called bimodal scoring (0-0-1-1) and the other is Likert scoring (0-1-2-3). The cut-off point limit for the bimodal scoring method is 2/3, and the maximum score that can be obtained is 12; for the Likert scale, it is 8/9, and the top score is 36.

The Perceived Stress Scale

The investigators used the Hungarian-language, validated version of the Perceived Stress Scale (PSS) to assess perceived stress. The questionnaire gives the investigators feedback on the stress level experienced during the past month. The questionnaire consists of 10 questions, which respondents can answer on a 5-point scale from 0-4, so the lowest possible score is 0, and the highest is 40. During the evaluation, based on the total scores, the respondents can be divided into 3 categories: 0-13 points = low level of perceived stress; 14-26 points = moderate perceived stress; 27-40 points = high level of perceived stress.

The International Physical Activity Questionnaire-Short Form

The investigators used the shortened version of the International Physical Activity Questionnaire (IPAQ-SF) to assess physical activity, validated in Hungarian. The questionnaire assesses the number of days and hours the subjects spend in heavy, moderate, or light physical work and examines the time all activities spent walking, lying down, and sitting for a period of one week.

The Premenstrual Assessment Form - Short Form

The investigators used the shortened version of the Premenstrual Assessment Form (PAF-SF), containing 10 questions translated into Hungarian to assess premenstrual symptoms. The questionnaire consists of 3 subscales; the first is called "Affect," which asks about increased irritability and bad mood, sad mood, stress, and overwork. The second subscale asks the participant about "Water retention," such as questions about edema and limb swelling, bloating, and weight gain. The third and last subscale assesses the existence of "Pain." It asks about lower abdominal cramps, back pain, joint pain, and pain caused by tense breasts. It is important to emphasize that all questions ask about the 7-14 days before menstruation and that the respondents can answer on a scale from one to six, the values of which are as follows: 1=uncharacteristic or no change; 2=minimal change; 3=slight change; 4=moderate change; 5=severe change; 6=very severe change. The total score can be calculated based on the scores given to these questions. The minimum number of points that can be obtained is 10, and the maximum number that can be obtained is 60. According to several international literature, the diagnostic point limit is 27, so this was used to evaluate the obtained data.

After evaluating the results of the PAF questionnaire, the investigators created a control and a case group to examine individual factors depending on the symptoms of PMS.

Among the applied statistical calculations, the minimum, maximum, mean (± standard deviation), and median (interquartile range) functions were used to characterize the descriptive statistics. During the normality test, the investigators used the Kolmogorov-Smirnov test, based on the results of which Spearman correlation analysis, independent sample T-test, Mann-Whitney U test, and Pearson chi-square test were performed to test the hypotheses.

The statistical data analysis software used in the study included Microsoft Excel 2016 and IBM SPSS version 28.0 (SPSS Inc., Chicago, IL, USA).

The level of significance was defined as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* women
* between the ages of 18-45 years
* regular menstruation

Exclusion Criteria:

* older than 45 years
* pregnancy
* amenorrhoea
* premature ovarian failure

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women between the ages of 18-45 who reported symptoms of PMS during the period of parameterization of the target group
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Premenstrual syndrome | 1 day
  * points;
  * Premenstrual Assessment Form Short Form Questionnaire (10 item version);
  * 1-6 point scale,
  * minimum score: 10 points;
  * maximum score: 60 points,
  * the higher the points the worse the symptoms

SECONDARY OUTCOMES:
Physical activity | 1 day
  minutes/week
Perceived Stress | 1 day
  * points;
  * Perceived Stress Scale;
  * 10 questions
  * 0-4 point scale,
  * minimum score: 0 points;
  * maximum score: 40 points,
  * the higher the points, the worse the symptoms:
  * 0-13 points: low level perceived stress
  * 14-26 points: medium level perceived stress
  * 27-40 points: high level perceived stress
Mental Health | 1 day
  * points;
  * General Health Questionnaire-12 items version;
  * 12 questions
  * 0-3 point scale,
  * two scoring methods: bimodal (0-0-1-1) and Likert-type (0-1-2-3).
  * the cut-off point for bimodal scoring is 3, and the maximum possible score is 12 points.
  * for Likert scoring, the maximum score is 36, and the cut-off point is 9.
BMI | 1 day
  kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Olívia Dózsa-Juhász, BSc, Study Chair — University of Pecs
Locations (1):
- University of Pécs, Pécs, Baranya, Hungary